CLINICAL TRIAL: NCT02171832
Title: Pharmacokinetics, Safety and Tolerability of a Single Dose of BI 1744 CL (20 μg Administered With the Respimat® Inhaler) in Patients With Mild and Moderate Hepatic Impairment (Child Pugh Classifications A and B) in Comparison to a Single Dose of BI 1744 CL (30 μg Administered With the Respimat® Inhaler) in Subjects With Normal Hepatic Function in a Monocentric, Open Label, Parallel Group Phase I Trial
Brief Title: Single Dose of BI 1744 CL in Patients With Mild and Moderate Hepatic Impairment Compared to Subjects With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1222.20
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy; Liver Diseases
MeSH Terms: conditions — Liver Diseases

ARMS (3):
- Mildly liver impaired patients (Experimental)
  Interventions: Drug: BI 1744 CL, low dose
- Moderately liver impaired patients (Experimental)
  Interventions: Drug: BI 1744 CL, low dose
- Healthy volunteers (Experimental)
  Interventions: Drug: BI 1744 CL, high dose

INTERVENTIONS:
Drug: BI 1744 CL, low dose
  Arms: Mildly liver impaired patients; Moderately liver impaired patients
Drug: BI 1744 CL, high dose
  Arms: Healthy volunteers

SUMMARY:
The main objective of this study was to investigate the influence of mild and moderate liver impairment on the pharmacokinetics, safety and selected pharmacodynamic parameters of BI 1744 CL in comparison to a control group with normal hepatic function after single orally inhaled administration of BI 1744 CL with the Respimat® Inhaler.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects:

* Healthy males and females according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests. The healthy subjects must meet the matching criteria based on the matching approach
* Age >21 and <75 years
* Body Mass Index (BMI) >18.5 and <32 kg/m2
* Creatinine clearance >70 mL/min according to Cockcroft & Gault
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Hepatically impaired subjects:

* Hepatically male and female impaired subjects determined by results of screening classified as

  * Group 1 (Child-Pugh A; Child-Pugh score of 5-6 points) and as
  * Group 2 (Child-Pugh B; Child-Pugh score of 7-9 points)
* Age >21 and <75 years
* BMI >18.5 and <34 kg/m2
* Creatinine clearance >40 mL/min according to Cockcroft & Gault (for hepatically impaired patients)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion Criteria:

Healthy subjects who meet any of the following criteria will not be entered into this trial:

* Any finding of the medical examination (including BP [>140 mmHg systolic and or >95 mmHg diastolic], PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Relevant gastrointestinal tract surgery (except appendectomy, herniotomy)
* Diseases of the central nervous system (such as epilepsy, seizures) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections (e.g. including Hepatitis B and C and HIV)
* History of allergy/hypersensitivity (including drug allergies) that are deemed relevant to the trial as judged by the investigator
* History or presence of allergy against iodine and/or contrast agent, latent or manifest hyperthyrosis or allergic diathesis to indocyanine green
* Intake of drugs that are contraindicated in connection with the indocyanine green test
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Participation in another trial with an investigational drug within one month after previous single dose administration or two months after previous multiple dose administration prior to administration or during the trial
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking when confined to the study site on trial days
* Alcohol abuse (more than 40 g/day in males, more than 20 g/day in females)
* Drug abuse, in the investigator's judgement upon review of the patient's history and urine screening for abused substances
* Veins unsuited for iv puncture on either arm (e.g. veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture)
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within 48 hours prior to trial or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance in the opinion of the investigator
* Inability to comply with dietary regimen of study centre
* Subjects not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions

Hepatically impaired subjects who meet any of the following criteria will not be entered into this trial:

* Medical disorder, condition or history of such that would impair the subject's ability to participate or complete this study in the opinion of the investigator or the sponsor
* Severe cerebrovascular or cardiac disorders, e.g. myocardial infarction less than 6 months prior to dosing, congestive heart failure of New York Heart Association (NYHA) grade III or IV, severe arrhythmia
* Relevant gastrointestinal tract surgery (except appendectomy, herniotomy, oesophagean varices)
* Diseases of the central nervous system (such as epilepsy, seizures) or psychiatric disorders or neurological disorders
* Evidence of hepatic encephalopathy related to chronic liver disease > grade 2 (exclusion by Number Connection Test)
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Resting heart rate in the awake subject below 45 beats per minute (BPM) or above 100 BPM; Systolic blood pressure below 100 mmHg or above 160 mmHg, Diastolic blood pressure above 95 mmHg
* Chronic or relevant acute infections (e.g. HIV) except e.g. Hepatitis B and C
* History of allergy/hypersensitivity (including drug allergies) that are deemed relevant to the trial as judged by the investigator
* History or presence of allergy against iodine and/or contrast agent, latent or manifest hyperthyrosis or allergic diathesis to indocyanine green
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial, excluded are those drugs, the patient is currently taking for treatment of the hepatic or concomitant disease.
* Change of chronic medication less than 4 weeks prior to dosing
* Participation in another trial with an investigational drug within one month after previous single dose administration or two months after previous multiple dose administration prior to administration or during the trial
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking when confined to the study site on trial days
* Alcohol abuse (more than 60 g/day in males, more than 40 g/day in females)
* Drug abuse, in the investigator's judgement upon review of the patient's history and urine screening for abused substances
* Veins unsuited for iv puncture on either arm (e.g. veins which are difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture)
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* History of Gastro intestinal tract bleeding within the past 3 months
* Excessive physical activities (within 48 hours prior to trial or during the trial)
* Clinically relevant laboratory abnormalities (except for liver function tests according to Child-Pugh classification or laboratory constellations of parameters that are typically altered in patients fulfilling the Child Pugh criteria) including relevant electrolyte disturbances
* Serum albumin <20 g/L
* Hemoglobin <8 g/dL
* Inability to comply with dietary regimen of study centre
* Subjects not able to understand and comply with protocol requirements, instructions and protocol-stated restrictions

Exclusion criteria specific for this study due to the known class side effect profile of ß2- mimetics (for healthy or hepatically impaired subjects):

* Asthma or history of pulmonary hyperreactivity
* Hyperthyrosis
* Allergic rhinitis in need of treatment
* Clinically relevant cardiac arrhythmia

For female subjects (healthy or hepatically impaired):

* Pregnancy or planning to become pregnant within 2 months of study completion
* Positive pregnancy test
* No adequate contraception in women of childbearing potential (adequate contraception: e.g. sterilisation, intrauterine device or oral contraception not containing ethinyl estradiol or ethinyl estradiol with an additional barrier method) for at least 3 months prior to participation in the study
* Inability to maintain this adequate contraception during the whole trial period.
* Lactation period

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
AUC0-∞,norm (dose-normalized area under the concentration time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | before and 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, and 72:00 hours following drug administration
Cmax,norm (dose-normalized maximum concentration of the analyte in plasma) | before and 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, and 72:00 hours following drug administration

SECONDARY OUTCOMES:
AUC0-∞ (area under the concentration time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | before and 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, and 72:00 hours following drug administration
Cmax (maximum concentration of the analyte in plasma) | before and 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, and 72:00 hours following drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | before and 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, and 72:00 hours following drug administration
AUC0-tz(,norm) ((dose-normalized ) area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | before and 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, and 72:00 hours following drug administration
%AUCtz-∞ (the percentage of the AUC 0-∞ that is obtained by extrapolation) | before and 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, and 72:00 hours following drug administration
λz (terminal rate constant in plasma) | before and 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, and 72:00 hours following drug administration
t1/2 (terminal half-life of the analyte in plasma) | before and 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, and 72:00 hours following drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | before and 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, and 72:00 hours following drug administration
MRTih (mean residence time of the analyte in plasma in the body after inhalation) | before and 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, and 72:00 hours following drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | before and 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, and 72:00 hours following drug administration
Aet1-t2 (amount of analyte that is eliminated in urine from the time point t1 to t2) | before and 0-8, 8-12, 12-24, 24-48, 48-72 hours following drug administration
fet1-t2 (fraction of analyte excreted in urine from the time point t1 to t2) | before and 0-8, 8-12, 12-24, 24-48, 48-72 hours following drug administration
CLR,t1-t2 (renal clearance of the analyte in urine from the time point t1 to t2) | before and 0-8, 8-12, 12-24, 24-48, 48-72 hours following drug administration
Plasma protein binding | before and 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, and 72:00 hours following drug administration
CL (total clearance of the analyte in plasma after intravascular administration) | before and 0:05, 0:10, 0:20, 0:40, 1:00, 2:00, 4:00, 6:00, 8:00, 12:00, 24:00, 48:00, and 72:00 hours following drug administration
Number of patients with abnormal findings in physical examination | Baseline, day 14
Number of patients with clinically significant changes in vital signs (blood pressure (BP), pulse rate (PR)) | Baseline, up to day 14
Number of patients with abnormal findings in 12-lead ECG (electrocardiogram) | Baseline, up to day 14
Number of patients with clinically significant changes in clinical laboratory tests | Baseline, up to day 14
Number of patients with adverse events | 5 weeks
Assessment of tolerability by the investigator on a 4-point scale | Day 14